CLINICAL TRIAL: NCT04885374
Title: China Amyotrophic Lateral Sclerosis Registry of Patients With Traditional Chinese Medicine
Acronym: CARE-TCM
Status: Recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, MD, PhD, Professor, Dongzhimen Hospital, Beijing
Other Study IDs: ALS-2021-CARE-TCM
Record Dates: First submitted 2021-05-08; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Amyotrophic lateral sclerosis patients: Amyotrophic lateral sclerosis patients with traditional Chinese medicine

SUMMARY:
A multi-center registration study of clinical characteristics of amyotrophic lateral sclerosis (ALS) patients with traditional Chinese medicine (TCM).

DETAILED DESCRIPTION:
The CARE-TCM is a prospective, multi-center, patient registry study. Eligible ALS patients with TCM treatments will be enrolled in the registry. After enrollment, this research collects the individual characteristics of patients' status. Longitudinal follow-up data are collected from both patients (primary caregivers) and their treating neurologists every 3 months for 5 years. The aims of the CARE-TCM are to: 1) explore the general characteristics of ALS patients with TCM and; 2) assess the effectiveness and safety of various TCMs on ALS based on nationwide registry outcome collecting process.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Patients with possible, laboratory supported probable, probable, or definite ALS according to the revised El Escorial criteria.
* ALS patients treated with traditional Chinese medicine.

Exclusion Criteria:

* Patients who refuse informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet the criteria will be enrolled from multi-centers in China.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Effective Survival | Through study completion, an average of 3 months
  The time from disease onset to death, tracheostomy, or permanent assisted ventilation

SECONDARY OUTCOMES:
Overall Survival | Through study completion, an average of 3 months
  Death owing to any causes
Rate of Disease Progression | Through study completion, an average of 3 months
  (48-total ALSFRS-R)/symptom duration (months)
Rate of Forced Vital Capacity (FVC) Decline | through study completion, an average of 3 months
  The slope of decline of forced vital capacity (FVC) to assess the respiratory function.
Rate of Body Mass Index (BMI) Decline | Through study completion, an average of 3 months
  The slope of decline of body mass index (BMI) to assess the disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, MD, PhD, Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital, Beijing University of Chinese Medicine, Beijing, China

REFERENCES:
- [Derived] Jia Q, Song Y, Zhang C, Li M, Feng L, Sugimoto K, Zhang X, Liu J, Gao Y. Reasons and experience for patients with amyotrophic lateral sclerosis using traditional Chinese medicine: a CARE-TCM based mixed method study. BMC Complement Med Ther. 2024 Jun 12;24(1):231. doi: 10.1186/s12906-024-04513-2. PMID 38867220
- [Derived] Song Y, Li M, Sugimoto K, Han Y, Liu J, Ma B, Song H, Zhang C, Gao Y; CARE-TCM Group. China amyotrophic lateral sclerosis registry of patients with Traditional Chinese Medicine (CARE-TCM): Rationale and design. J Ethnopharmacol. 2022 Feb 10;284:114774. doi: 10.1016/j.jep.2021.114774. Epub 2021 Oct 23. PMID 34699945